CLINICAL TRIAL: NCT06037694
Title: Widening of Keratinized Tissues With an Expanded Meshed Free Gingival Graft: a Multi-center Randomized Controlled Trial.
Brief Title: Effectiveness of Meshed Free Gingival Graft for Widening of Keratinized Tissues
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OCarcuac-meshFGG
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2024-10

CONDITIONS: Gingiva Atrophy
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Free Gingival Graft (Active Comparator): A mucogingival surgery where a conventional free gingival graft harvested from the palate is placed on a recipient site prepared to increase the width of KM at implant sites.
  Interventions: Procedure: Conventional Free Gingival Graft
- Meshed Free Gingival Graft (Experimental): A mucogingival surgery where a meshed free gingival graft harvested from the palate is placed on a recipient site prepared to increase the width of KM at implant sites.
  Interventions: Procedure: 'Mesh Free Gingival Graft

INTERVENTIONS:
Procedure: Conventional Free Gingival Graft — Implant site with insufficient dimensions of KM will be covered by a conventional free gingival graft.
  Arms: Free Gingival Graft
Procedure: 'Mesh Free Gingival Graft — Implant site with insufficient dimensions of KM will be covered by a expanded meshed free gingival graft.
  Arms: Meshed Free Gingival Graft

SUMMARY:
The overall objective of this project is to evaluate, over a period of 1 year, the outcomes of either conventional free gingival graft (FGG) or mesh-FGG to increase the width of keratinized mucosa (KM) at implant sites.

DETAILED DESCRIPTION:
The importance of the width of keratinized mucosa (KM) at implant sites remains a subject of ongoing debate. Reduced dimensions of KM (width <2 mm) are associated with mucosal recession, biofilm accumulation, soft-tissue inflammation, marginal bone loss, peri-implantitis and patient discomfort. Surgical options to increase the width of KM include an apically positioned flap, either alone or in combination with an autogenous graft or a xenogeneic collagen matrix. The free gingival graft (FGG) is a well-established technique with a history of successful clinical use. The harvesting procedure for autogenous graft from the palatal mucosa, however, is usually associated with significant patient morbidity, especially when there is a need to graft extensive mucosal areas. To overcome this problem, various graft modifications have been proposed to limit the need for large-area autografts. Examples include the accordion technique, the strip gingival autograft technique, and a vertical modification of the strip gingival graft. The expanded mesh graft, another graft modification, has been used in the field of plastic surgery, especially in the treatment of large burn wounds. Recently, De Greef, Carcuac, De Mars et al. proposed this technique to be used in periodontal plastic surgery, more specifically, in the widening of KM at implant sites by means of a meshed free gingival graft (mesh-FGG). In this case series, initially inadequate width of KM in edentulous areas could be successfully increased prior to implant installation, without the need for any extensive autograft harvesting. Data from trials comparing mesh-FGG to conventional FGG and assessing the long-term efficacy of this novel technique, however, are missing.

The investigators hypothesize that the mesh-FGG technique will demonstrate similar clinical results (non-inferiority: increase in KM width) but improved patient-reported outcomes (superiority: post-surgical morbidity) compared to the FGG.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age,
* systemically healthy,
* presence of ≥2 adjacent implants in both sides of the mandibles showing <2 mm of KM on the buccal aspects,
* subjects have to present with discomfort from brushing and/or difficulties in maintaining proper home care due to inadequate dimension of KM
* Full-Mouth Plaque Score (FMPS) <20%,
* Full-Mouth Bleeding Score (FMBS) <20%.

Exclusion Criteria:

* pregnancy or lactation,
* tobacco smoking,
* uncontrolled medical condition,
* medication that can affect gingival conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Keratinized Mucosa width (KMW) | up to 1 year
  Measured as the distance from the muco-gingival-junction to the occlusal portion of the mucosa

SECONDARY OUTCOMES:
Changes of Keratinized Mucosa Thickness (KMT) | up to 1 year
  measured by a therapeutic probe with a rubber stop
Patient Morbidity | up to 2 weeks
  Measured with Visual Analogue Scale (VAS), which consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Patient Satisfaction | up to 1 year
  Measured with Visual Analogue Scale (VAS), which consists of a 10cm line, with two end points representing 0 ('not satisfied') and 10 ('satisfied as much as it could possibly be')

CONTACTS AND LOCATIONS:
Overall Officials: Jan Derks, Study Chair — Goteborg University
Locations (1):
- ConfiDent ® Dental Surgery Clinic, Dubai Palm Jumeirah, Dubai, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Clin Periodontol. 2018 Jun;45 Suppl 20:S246-S266. doi: 10.1111/jcpe.12954. PMID 29926484
- [Background] Sanz M, Schwarz F, Herrera D, McClain P, Figuero E, Molina A, Monje A, Montero E, Pascual A, Ramanauskaite A, Renouard F, Sader R, Schiegnitz E, Urban I, Heitz-Mayfield L. Importance of keratinized mucosa around dental implants: Consensus report of group 1 of the DGI/SEPA/Osteology Workshop. Clin Oral Implants Res. 2022 Jun;33 Suppl 23:47-55. doi: 10.1111/clr.13956. PMID 35763021
- [Background] Lim HC, An SC, Lee DW. A retrospective comparison of three modalities for vestibuloplasty in the posterior mandible: apically positioned flap only vs. free gingival graft vs. collagen matrix. Clin Oral Investig. 2018 Jun;22(5):2121-2128. doi: 10.1007/s00784-017-2320-y. Epub 2017 Dec 23. PMID 29275490
- [Background] Tavelli L, Barootchi S, Avila-Ortiz G, Urban IA, Giannobile WV, Wang HL. Peri-implant soft tissue phenotype modification and its impact on peri-implant health: A systematic review and network meta-analysis. J Periodontol. 2021 Jan;92(1):21-44. doi: 10.1002/JPER.19-0716. Epub 2020 Aug 9. PMID 32710810
- [Background] Singh M, Nuutila K, Collins KC, Huang A. Evolution of skin grafting for treatment of burns: Reverdin pinch grafting to Tanner mesh grafting and beyond. Burns. 2017 Sep;43(6):1149-1154. doi: 10.1016/j.burns.2017.01.015. Epub 2017 Jan 30. PMID 28153583
- [Background] De Greef A, Carcuac O, De Mars G, Stankov V, Cortasse B, Giordani G, Van Dooren E. The expanded mesh free gingival graft: A novel approach to increase the width of keratinized mucosa. Clin Adv Periodontics. 2024 Sep;14(3):157-164. doi: 10.1002/cap.10264. Epub 2023 Aug 16. PMID 37551510
- [Background] Thoma DS, Naenni N, Figuero E, Hammerle CHF, Schwarz F, Jung RE, Sanz-Sanchez I. Effects of soft tissue augmentation procedures on peri-implant health or disease: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Mar;29 Suppl 15:32-49. doi: 10.1111/clr.13114. PMID 29498129